CLINICAL TRIAL: NCT06479616
Title: A Long-term Follow-up Study Evaluating the Safety and Efficacy of Subjects With β-thalassemia Treated With Base-edited Autologous Hematopoietic Stem Cell (CS-101) Transplantation
Brief Title: A Long-term Follow-up Study in Participants Who Received CS-101
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CS-101-04
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- long term follow up (Experimental): All participants who complete CS-101-03(NCT0606518) studie after CS-101 infusion will be asked to participate in this long-term follow-up study.
  Interventions: Genetic: CS-101

INTERVENTIONS:
Genetic: CS-101 — Autologous CD34+ hematopoietic stem cell suspension modified by in vitro base editing technique

SUMMARY:
This is a study to evaluate the long-term safety and efficacy of CS-101 in participants who received CS-101 in study CS -101-03 (NCT06065189)

DETAILED DESCRIPTION:
This is a study to evaluate the long-term safety and efficacy of CS-101 in participants who received CS-101 in study CS -101-03 (NCT06065189) .

Subjects in the CS-101-03 study will be entered into long-term follow-up of this study up to 2 years post-infusion at the completion of the last (6-month) follow-up visit after treatment with CS-101 Injection.

ELIGIBILITY:
Inclusion Criteria:

* Participants (or his or her legally appointed and authorized representative or guardian) must sign and date informed consent form (ICF) and, where applicable, an assent form
* Participants must have received CS-101 infusion in last IIT study

Exclusion Criteria:

* There are no exclusion criteria

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of SAEs and CS-101 related AES as assessed by CTCAE v5.0 | Signing of informed consent up to 2 years post CS-101 infusion
  CommonTerminology Criteria for Adverse Events（CTCAE）has 5 levels of AE determination, increasing in severity as the level increases
Occurrence of all-cause death | Signing of informed consent up to 2 years post CS-101 infusion
New malignancies and hematologic disorders | Signing of informed consent up to 2 years post CS-101 infusion
  Based on ICD-11
Occurrence of achieving transfusion independence for at least 12 consecutive months | From 3 months after last RBC transfusion up to 2 years post CS-101 infusion

SECONDARY OUTCOMES:
Change in fetal hemoglobin(HbF) concentration over time | up to 2 years post-CS-101 infusion
Change in total hemoglobin(Hb) concentration over time | up to 2 years post-CS-101 infusion
Chimerism level in Peripheral blood and bone marrow Proportion of alleles with intended genetic modification in peripheral blood leukocytes and bone marrow over time | up to 2 years post-CS-101 infusion
  Proportion of alleles with intended genetic modification in peripheral blood leukocytes and bone marrow over time

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Zhai, M.D., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China